CLINICAL TRIAL: NCT01788150
Title: Direct Implantation of Rapamycin-Eluting Stents With Bio-Erodible Drug Carrier Technology Utilizing the Second Generation Svelte Drug-Eluting Coronary Stent Integrated Delivery System (IDS)
Brief Title: Safety and Efficacy Study of the Svelte Drug-Eluting Coronary Stent Delivery System
Acronym: DIRECT II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Svelte Medical Systems, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IP-12-002
Record Dates: First submitted 2013-02-05; First posted 2013-02-11 (Estimated); Results first posted 2021-05-04 (Actual); Last update posted 2021-05-04 (Actual); Status verified 2021-04

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Svelte Drug-Eluting Coronary Stent (Experimental): Coronary Stenting
  Interventions: Device: Coronary Stenting
- Medtronic Resolute Integrity Drug-Eluting Stent (Active Comparator): Coronary Stenting
  Interventions: Device: Coronary Stenting

INTERVENTIONS:
Device: Coronary Stenting

SUMMARY:
A prospective, randomized, active-control, multi-center clinical trial comparing the safety and efficacy of the Svelte Drug-Eluting Coronary Stent Integrated Delivery System (IDS) to that of the commercially available Resolute IntegrityTM Drug-Eluting Stent.

The study objective is to assess the safety and efficacy of the Svelte Drug-Eluting Coronary Stent Integrated Delivery System (IDS) compared to the Resolute IntegrityTM Drug-Eluting Stent in patients with single, never previously treated coronary artery lesions

ELIGIBILITY:
Inclusion Criteria:

General Inclusion Criteria

1. Patient is ≥18 years old;
2. Patient is eligible for percutaneous coronary intervention (PCI);
3. Patient is an acceptable candidate for emergent coronary artery bypass graft (CABG) surgery;
4. Patient has clinical evidence of ischemic heart disease, stable or unstable angina, silent ischemia, or a positive functional study;
5. Female subjects of childbearing potential must have a negative pregnancy test within 7-days before the trial procedure;
6. Patient or subject's legal representative has been informed of the nature of the trial and agrees to its provisions and has provided written informed consent as approved by the Hospital Research Ethics Committee (HREC) of the respective investigational site; and
7. Patient agrees to comply with specified follow-up evaluations and to return to the same investigational site where the procedure was performed.

Angiographic Inclusion Criteria

1. Patient has either a single target lesion, or two lesions (target and non-target) located in separate coronary arteries;
2. If a non-target lesion is treated, it must be treated first and only with commercially available PTCA balloons and/or stents. Post PCI of the non-target vessel, all of the following conditions must be met:

   1. Residual diameter stenosis < 30%;
   2. Absence of any angiographic complications;
   3. Absence of ischemic symptoms; and
   4. Absence of significant new arrhythmia or ECG monitoring changes suggestive of ischemia.
3. Reference vessel ≥ 2.5 mm and ≤ 3.5 mm in diameter by visual estimate;
4. Target lesion < 20 mm in length by visual estimate (the intention is to cover the entire lesion with one stent of adequate length); and
5. Target lesion stenosis ≥ 50% and < 100% by visual estimate.

Exclusion Criteria:

General Exclusion Criteria

1. Patient is currently enrolled in another investigational device or drug trial that has not completed the primary endpoint or that clinically interferes with the current study endpoints Note: Trials requiring extended follow-up for products that were investigational, but have since become commercially available, are not considered investigational trials;
2. The patient requires a staged procedure of the target vessel within 6-months or a staged procedure of a non-target vessel within 30-days post-procedure;
3. The target lesion requires treatment with a device other than PTCA prior to stent placement (such as, but not limited to, directional coronary atherectomy, excimer laser, rotational atherectomy, etc.);
4. Any DES deployment anywhere in the target vessel within the past 9-months;
5. Any BMS deployment anywhere in the target vessel within the past 6-months;
6. Any previous stent placement within 10 mm (proximal or distal) of the target lesion;
7. Myocardial infarction within 72-hours of the index procedure, with the exception of:

   1. Patients who have had a STEMI and PCI to the culprit lesion may be included if they have a suitable lesion in another vessel, and have been clinically and hemodynamically stable for 72-hours;
   2. Patients who have had a non-STEMI may be included if their troponin levels are within the laboratory normal range within 24-hours pre-procedure.
8. Co-morbid condition(s) that could limit the patient's ability to participate in the trial or to comply with follow-up requirements, or impact the scientific integrity of the trial;
9. Concurrent medical condition with a life expectancy of less than 12-months;
10. Documented left ventricular ejection fraction (LVEF) ≤ 30%;
11. Unstable angina pectoris from an extra-cardiac cause (Braunwald Class A I-III);
12. Known allergies to the following: Acetylsalicylic acid (ASA), Clopidogrel bisulfate, Ticlopidine, Prasugrel, Rapamycin, Zotarolimus, PEAIII AcBz, Heparin/ Bivalirudin, or contrast agent (that cannot be adequately premedicated);
13. Platelet count < 100,000 cells/mm3 or > 700,000 cells/mm3 or a WBC < 3.000 cells/mm3 or hemoglobin < 100g/l;
14. Acute or chronic renal dysfunction (serum creatinine > 170μmol/L);
15. History of a stroke or transient ischemic attack (TIA) within the prior 6-months;
16. Active peptic ulcer or upper gastrointestinal (GI) bleeding within the prior 6-months;
17. History of bleeding diathesis or coagulopathy or will refuse blood transfusions; and
18. Patients requiring ongoing anticoagulation with warfarin or dabigatran.

Angiographic Exclusion Criteria

1. Total occlusion (TIMI 0 or 1);
2. Target vessel has angiographic evidence of thrombus
3. Target vessel is excessively tortuous or has heavy calcification;
4. Significant (> 50%) stenosis proximal or distal to the target lesion that might require revascularization or impede run off;
5. Target lesion is located in or supplied by an arterial or venous bypass graft;
6. Ostial target lesion (within 5.0 mm of vessel origin) or any location within the left main coronary artery;
7. Target lesion involves a side branch > 2.0 mm in diameter; and
8. Unprotected Left Main coronary disease (stenosis > 50%).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2014-05 (Actual); Study Completion 2019-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Verheye, MD, PhD, Principal Investigator — Antwerp Cardiovascular Institute; Alexandre Abizaid, MD, PhD, Principal Investigator — Instituto Dante Pazzanese de Cardiologia
Locations (18):
- Belgium (4):
  - OLV Ziekenhuis Aalst, Aalst
  - Middelheim Ziekenhuis, Antwerp
  - ZOL Genk, Genk
  - CHU Liège, Liège
- Všeobecná fakultní nemocnice Praha, Prague, Czechia
- France (3):
  - Clinique Saint-Hilaire, Rouen
  - CHU de Toulouse, Toulouse
  - Clinique Pasteur, Toulouse
- Germany (2):
  - Medizinisches Verzorgungszentrum Prof. Mathey, Prof. Schofer, Hamburg
  - University Medical Center Hamburg-Eppendorf, Hamburg
- Netherlands (5):
  - OLVG Amsterdam, Amsterdam
  - Catharina Hospital Eindhoven, Eindhoven
  - Erasmus MC, Rotterdam
  - Maasstad Ziekenhuis, Rotterdam
  - University Medical Center Utrecht, Department of Cardiology, Utrecht
- Sweden (2):
  - Skane University Hospital, Malmo
  - Södersjukhuset, Stockholm
- Inselspital, Bern, Switzerland

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Svelte Drug-Eluting Coronary Stent | Medtronic Resolute Integrity Drug-Eluting Stent
Started | 108 | 51
Completed | 95 | 48
Not Completed | 13 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Svelte Drug-Eluting Coronary Stent | Medtronic Resolute Integrity Drug-Eluting Stent | Total
Number analyzed (Participants) | 108 | 51 | 159
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.7 (9.9) | 64.2 (12.4) | 63.2 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 17 | 43
  Male | 82 | 34 | 116
Region of Enrollment [Number; unit: participants]
  Netherlands | 33 | 20 | 53
  Sweden | 1 | 1 | 2
  Belgium | 24 | 16 | 40
  Czechia | 3 | 5 | 8
  France | 26 | 6 | 32
  Switzerland | 14 | 2 | 16
  Germany | 7 | 1 | 8

OUTCOME MEASURES:

1. Primary Outcome: Angiographic In-Stent Late Lumen Loss (LL)
Description: Defined as the measurements either within the stented segment or within 5 mm proximal and distal to the stent edges.
Time Frame: 6-months post-procedure
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Svelte Drug-Eluting Coronary Stent | Medtronic Resolute Integrity Drug-Eluting Stent
Number analyzed (Participants) | 89 | 40
mm | 0.09 (0.31) | 0.13 (0.27)

2. Secondary Outcome: Number of Participants Clinically-driven Target Lesion Revascularization (TLR)
Description: Clinically driven TLR is defined as revascularization performed on a patient who returns with clinical symptoms such as unstable angina, that is, chest pain that increases in frequency, intensity or duration.
Time Frame: 1 year post-procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Svelte Drug-Eluting Coronary Stent | Medtronic Resolute Integrity Drug-Eluting Stent
Number analyzed (Participants) | 108 | 51
Participants | 2 | 1

3. Secondary Outcome: Number of Participants Composite of Cardiac Death, MI Attributed to the Target Vessel and Clinically Driven Target Lesion Revascularization
Description: Composite of cardiac death, MI attributed to the target vessel and clinically driven target lesion revascularization
Time Frame: 1 year post-procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Svelte Drug-Eluting Coronary Stent | Medtronic Resolute Integrity Drug-Eluting Stent
Number analyzed (Participants) | 108 | 51
Participants | 4 | 4

4. Secondary Outcome: Number of Participants Composite of All-cause Mortality, Any MI and Any Revascularization, Target Vessel Revascularization or Revascularization of Non Target Vessels
Description: Composite of all-cause mortality, any MI and any revascularization, target vessel revascularization or revascularization of non target vessels
Time Frame: 1 year post-procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Svelte Drug-Eluting Coronary Stent | Medtronic Resolute Integrity Drug-Eluting Stent
Number analyzed (Participants) | 108 | 51
Participants | 18 | 9

5. Secondary Outcome: Number of Participants Stent Thrombosis
Description: The sudden occlusion of a stented coronary artery due to thrombus formation.
Time Frame: 1 year post-procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Svelte Drug-Eluting Coronary Stent | Medtronic Resolute Integrity Drug-Eluting Stent
Number analyzed (Participants) | 108 | 51
Participants | 0 | 0

6. Secondary Outcome: Number of Participants Acute Success Rates
Description: Direct Stenting Success, Lesion Success, Procedure Success and Device Failure
Time Frame: From index procedure to hospital discharge, an average of 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Svelte Drug-Eluting Coronary Stent | Medtronic Resolute Integrity Drug-Eluting Stent
Number analyzed (Participants) | 108 | 51
Participants
  Device Failure | 2 | 0
  Direct Stenting Success | 96 | 45
  Lesion Success | 104 | 51
  Procedure Success | 103 | 48

7. Secondary Outcome: Number of Participants In-stent and In-segment Angiographic Binary Restenosis Rate
Description: The rate which restenosis occurs
Time Frame: 6-months post-procedure
Population: 19 Subjects in the Svelte Arm and 11 subjects in the Medtronic Arm did not return for their 6 month follow-up or refused to have the invasive follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Svelte Drug-Eluting Coronary Stent | Medtronic Resolute Integrity Drug-Eluting Stent
Number analyzed (Participants) | 89 | 40
Participants
  In-stent angiographic binary restenosis rate | 2 | 0
  In-segment angiographic binary restenosis rate | 5 | 0

8. Secondary Outcome: In-stent and In-segment Minimum Lumen Diameter
Description: Smallest diameter in the stent or segment area
Time Frame: 6-months post-procedure
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Svelte Drug-Eluting Coronary Stent | Medtronic Resolute Integrity Drug-Eluting Stent
Number analyzed (Participants) | 89 | 40
mm
  In-stent minimum lumen diameter | 2.28 (0.46) | 2.52 (0.45)
  In-segment minimum lumen diameter | 2.07 (0.48) | 2.26 (0.48)

9. Secondary Outcome: In-segment Late Lumen Loss
Description: Late lumen loss is the difference in millimeters between the diameter of a stented segment post-procedure compared with the follow-up angiogram
Time Frame: 6-months post-procedure
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Svelte Drug-Eluting Coronary Stent | Medtronic Resolute Integrity Drug-Eluting Stent
Number analyzed (Participants) | 89 | 40
mm | 0.04 (0.33) | -0.02 (0.30)

10. Secondary Outcome: Neointimal Hyperplasia as Measured by OCT
Description: (% lumen volume)
Time Frame: 6-months post procedures
Population: 8 Subjects in the Svelte Arm refused to have the follow-up OCT at 6 months. This was only measureed in the Svelte arm.
Measure: Mean (Standard Deviation); unit: percentage of lumen volume
Arm/Group | Svelte Drug-Eluting Coronary Stent
Number analyzed (Participants) | 22
percentage of lumen volume | 11.3 (4.7)

11. Secondary Outcome: Strut Coverage
Description: (% of struts malapposed, protruding non-covered, protruding covered, non-protruding covered)
Time Frame: 6-months post procedure
Population: 8 Subjects in the Svelte Arm refused to have the follow-up OCT at 6 months. This was only measured int he Svelte arm
Measure: Mean (Standard Deviation); unit: % strut coverage
Arm/Group | Svelte Drug-Eluting Coronary Stent
Number analyzed (Participants) | 22
% strut coverage | 94.2 (9.0)

12. Secondary Outcome: Number of Participants Target Vessel Failure
Description: Composite endpoint of cardiac death, target vessel MI (Q or Non-Q wave), or clinically- driven target vessel revascularization (TVR) by percutaneous or surgical methods.
Time Frame: 1 year post procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Svelte Drug-Eluting Coronary Stent | Medtronic Resolute Integrity Drug-Eluting Stent
Number analyzed (Participants) | 108 | 51
Participants | 7 | 5

ADVERSE EVENTS:
Arm/Group | Svelte Drug-Eluting Coronary Stent | Medtronic Resolute Integrity Drug-Eluting Stent
All-Cause Mortality (participants affected / at risk) | 0/108 | 0/51
Serious Adverse Events (participants affected / at risk) | 21/108 | 8/51
Other Adverse Events (participants affected / at risk) | 36/108 | 14/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Svelte Drug-Eluting Coronary Stent (N=108) | Medtronic Resolute Integrity Drug-Eluting Stent (N=51)
Angina (Cardiac disorders) | 2 (2) | 0 (0)
Arrhythmia (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac decompensation (Cardiac disorders) | 1 (1) | 0 (0)
HYperthyroidism (Endocrine disorders) | 1 (1) | 0 (0)
GI Bleed (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Local Infection (Infections and infestations) | 0 (0) | 2 (2)
Depression (Nervous system disorders) | 1 (1) | 0 (0)
Fainting/Syncope/Vasovagal Reaction (Nervous system disorders) | 0 (0) | 1 (1)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Other respiratory (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Renal Failure/Insufficiency (Renal and urinary disorders) | 0 (0) | 1 (1)
Atypical Chest Pain (General disorders) | 1 (1) | 1 (1)
Fever/Pyrexia (Immune system disorders) | 1 (1) | 0 (0)
Chest pain wihtout cardiac enzyme elevation (General disorders) | 1 (1) | 0 (0)
Endometrium Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Black-out after drinking wine (General disorders) | 1 (1) | 0 (0)
Carotid Stenosis (Vascular disorders) | 1 (1) | 0 (0)
Silent Ischemia (Cardiac disorders) | 1 (1) | 0 (0)
Claudication (Vascular disorders) | 2 (2) | 0 (0)
Restenosis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Svelte Drug-Eluting Coronary Stent (N=108) | Medtronic Resolute Integrity Drug-Eluting Stent (N=51)
MI (Cardiac disorders) | 13 (13) | 11 (11)
Elevated cardiac enzymes (Cardiac disorders) | 8 (8) | 3 (3)
Dissection (Vascular disorders) | 9 (9) | 0 (0)
Atypical Chest pain (General disorders) | 6 (6) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No